CLINICAL TRIAL: NCT02858440
Title: Immunogenicity and Safety of GSK Biologicals' Combined Diphtheria-tetanus-acellular Pertussis-inactivated Poliovirus and Haemophilus Influenzae Type b (DTPa-IPV/Hib) Conjugate Vaccine
Brief Title: A Study to Assess the Immunogenicity and Safety of GSK Biologicals' Infanrix-IPV/Hib Vaccine Administered as a Three-dose Vaccination Course at 3, 4.5 and 6 Months of Age and a Booster Dose at 18 Months of Age in Healthy Infants in Russia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116194; 2013-005577-43 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type b
Keywords: Primary dose; Reactogenicity; Immunogenicity; Booster dose; Combined vaccine; Russian Infants; Infanrix®-IPV/Hib
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (1):
- DTPa-IPV/Hib Group (Experimental): All subjects receive three doses of primary vaccination of the study vaccine, Infanrix-IPV/Hib (DTPa-IPV/Hib), at 3, 4.5 and 6 months of age and a single dose of booster vaccination at 18 months of age. The vaccine is administered intramuscularly into the upper side of the thigh on the right/left side.
  Interventions: Biological: Infanrix-IPV/Hib

INTERVENTIONS:
Biological: Infanrix-IPV/Hib — Subjects receive Infanrix-IPV/Hib three-dose primary vaccination course at 3, 4.5 and 6 months of age and a booster dose at 18 months of age. The vaccine is administered intramuscularly into the upper side of the thigh on the right/left side.

SUMMARY:
The purpose of this study is to evaluate the immune response, safety and reactogenicity after receiving combined DTPa-IPV/Hib vaccine when administered as a three-dose primary vaccination course at 3, 4.5 and 6 months of age and as a booster dose at 18 months of age in Russian healthy children according to the Russian immunisation schedule

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representatives [LARs] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female child between 3 and 4 months of age at the time of the first vaccination.
* Written informed consent obtained from the parents/LARs of the subject prior to performing any study specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting since birth. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of hepatitis B and other vaccines given as part of the national immunisation schedule and as part of routine vaccination practice, that are allowed at any time during the study period. Seasonal or pandemic influenza vaccine can be given at any time during the study, and according to the Summary of Product Characteristics and national recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis and Hib diseases.
* History of diphtheria, tetanus, pertussis, poliomyelitis and Hib diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects.
* Serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C for oral, axillary or tympanic route, or ≥38.0°C for rectal route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 3 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Russia (5):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Romanenko V, Osipova I, Galustyan A, Scherbakov M, Baudson N, Farhi D, Anaya L, Kuriyakose SO, Meyer N, Janssens W. Immunogenicity and safety of a combined DTPa-IPV/Hib vaccine administered as a three-dose primary vaccination course and a booster dose in healthy children in Russia: a phase III, non-randomized, open-label study. Hum Vaccin Immunother. 2020 Sep 1;16(9):2265-2273. doi: 10.1080/21645515.2020.1720437. Epub 2020 Feb 12. PMID 32048889

RESULTS

PARTICIPANT FLOW:
Groups:
- DTPa-IPV/Hib Group: All subjects received three doses of primary vaccination of the study vaccine, Infanrix-IPV/Hib (DTPa-IPV/Hib), at 3, 4.5 and 6 months of age and a single dose of booster vaccination at 18 months of age. The vaccine was administered intramuscularly into the upper side of the thigh on the right/left side.
Period: Overall Study
Arm/Group | DTPa-IPV/Hib Group
Started | 235
Completed | 223
Not Completed | 12
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 2
Not completed — Consent withdrawal | 3
Not completed — Migrated/moved from study area | 4

BASELINE CHARACTERISTICS:
Groups:
- DTPa-IPV/Hib Group: All subjects received three doses of primary vaccination of the study vaccine, DTPa-IPV/Hib, at 3, 4.5 and 6 months of age and a single dose of booster vaccination at 18 months of age. The vaccine was administered intramuscularly into the upper side of the thigh on the right/left side.
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 235
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 14.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 235

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T), Post Primary Vaccination
Description: A seroprotected subject is a subject whose anti-D and anti-T antibody concentration was greater than or equal to (≥) 0.1 International Units per milliliter (IU/mL).
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: The According-to-protocol (ATP) cohort for analysis of immunogenicity of the primary epoch included all evaluable subjects who complied with protocol and for whom assay results were available for antibodies against at least one study vaccine antigen component one month after Dose 3.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
Participants
  Anti-D antibody ≥ 0.1 IU/mL | 176
  Anti-T antibody ≥ 0.1 IU/mL | 176

2. Primary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Types 1, 2 and 3, Post Primary Vaccination
Description: A seroprotected subject is a subject whose anti-poliovirus types 1, 2 and 3 antibody titer was ≥ 8 ED50.
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 151
Participants
  Anti-Polio 1 antibody ≥ 8 ED50 | 151
  Anti-Polio 2 antibody ≥ 8 ED50 | 151
  Anti-Polio 3 antibody ≥ 8 ED50 | 150

3. Primary Outcome: Number of Seroprotected Subjects for Anti-polyribosyl Ribitol Phosphate (Anti-PRP), Post Primary Vaccination
Description: A seroprotected subject is a subject whose anti-PRP antibody concentration was ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 182
Participants | 179

4. Primary Outcome: Number of Seropositive Subjects for Anti-pertussis (Anti- PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN), Post Primary Vaccination
Description: A seropositive subject is a subject whose antibody concentration was ≥ 2.046 IU/mL for anti-FHA, ≥ 2.187 IU/mL for anti-PRN and ≥ 2.693 IU/mL for anti-PT.
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
Participants
  Anti-FHA antibody ≥ 2.046 IU/mL | 175
  Anti-PRN antibody ≥ 2.187 IU/mL | 175
  Anti-PT antibody ≥ 2.693 IU/mL | 174

5. Secondary Outcome: Number of Seroprotected Subjects for Anti-D and Anti-T, Post Booster Vaccination
Description: A seroprotected subject is a subject whose anti-D and anti-T antibody concentration was ≥ 0.1 IU/mL.
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: The ATP cohort for analysis of immunogenicity of the booster epoch included all evaluable subjects who complied with protocol and for whom assay results were available for antibodies against at least one study vaccine antigen component one month after the booster dose.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
Participants
  anti-D antibody | 188
  anti-T antibody | 188

6. Secondary Outcome: Number of Seroprotected Subjects for Anti-poliovirus Types 1, 2 and 3, Post Booster Vaccination
Description: A seroprotected subject is a subject whose anti-poliovirus types 1, 2 and 3 antibody titer was ≥ 8 ED50.
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
Participants
  anti-Polio 1 antibody | 176
  anti-Polio 2 antibody: number analyzed (Participants) | 169
  anti-Polio 2 antibody | 169
  anti-Polio 3 antibody: number analyzed (Participants) | 167
  anti-Polio 3 antibody | 167

7. Secondary Outcome: Number of Seroprotected Subjects for Anti-PRP, Post Booster Vaccination
Description: A seroprotected subject is a subject whose anti-PRP antibody concentration was ≥ 0.15 µg/mL.
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
Participants | 188

8. Secondary Outcome: Number of Seropositive Subjects for Anti- PT, Anti-FHA and Anti-PRN, Post Booster Vaccination
Description: as for outcome 4
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
Participants
  anti-PT antibody | 188
  anti-FHA antibody | 188
  anti-PRN antibody: number analyzed (Participants) | 187
  anti-PRN antibody | 187

9. Secondary Outcome: Antibody Concentrations for Anti-D and Anti-T, Post Primary Vaccination
Description: The antibody concentrations for anti-D and anti-T were presented as geometric mean concentrations (GMCs) and expressed as IU/mL.
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
IU/mL
  Anti-D antibody | 3.24 [2.84 to 3.68]
  Anti-T antibody | 3.14 [2.81 to 3.51]

10. Secondary Outcome: Antibody Concentrations for Anti-D and Anti-T, Post Booster Vaccination
Description: as for outcome 9
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
IU/mL
  anti-D antibody | 12.11 [10.82 to 13.56]
  anti-T antibody | 8.18 [7.35 to 9.11]

11. Secondary Outcome: Antibody Titers for Anti-polio Types 1, 2 and 3, Post Primary Vaccination
Description: The antibody titers for anti-polio types 1, 2 and 3 were presented as geometric mean titres (GMTs).
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 151
Titers
  Anti-Polio 1 antibody | 613.9 [505.5 to 745.5]
  Anti-Polio 2 antibody | 591.6 [487.3 to 718.3]
  Anti-Polio 3 antibody | 827.4 [674.7 to 1014.6]

12. Secondary Outcome: Antibody Titers for Anti-polio Types 1, 2 and 3, Post Booster Vaccination
Description: The antibody titers for anti-polio types 1, 2 and 3 were presented as geometric mean titres (GMTs).
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
Titers
  anti-Polio 1 antibody | 2185.4 [1901.1 to 2512.3]
  anti-Polio 2 antibody: number analyzed (Participants) | 169
  anti-Polio 2 antibody | 2944.1 [2601.3 to 3332.2]
  anti-Polio 3 antibody: number analyzed (Participants) | 167
  anti-Polio 3 antibody | 3684.6 [3225.3 to 4209.3]

13. Secondary Outcome: Antibody Concentration for Anti-PRP, Post Primary Vaccination
Description: The antibody concentrations for anti-PRP were presented as geometric mean concentrations (GMCs) and expressed as µg/mL.
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 182
µg/mL | 2.97 [2.48 to 3.54]

14. Secondary Outcome: Antibody Concentration for Anti-PRP, Post Booster Vaccination
Description: The antibody concentrations for anti-PRP were presented as geometric mean concentrations (GMCs) and expressed as µg/mL.
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
µg/mL | 28.72 [24.70 to 33.40]

15. Secondary Outcome: Antibody Concentrations for Anti-PT, Anti-FHA and Anti-PRN, Post Primary Vaccination
Description: The antibody concentrations for anti-PT, anti-FHA and anti-PRN were presented as GMCs and expressed as IU/mL.
Time Frame: At Month 4 (i.e. one month after 3rd dose of primary vaccination)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 176
IU/mL
  Anti-FHA antibody | 120.2 [107.0 to 135.1]
  Anti-PRN antibody | 166.1 [146.8 to 187.8]
  Anti-PT antibody | 65.0 [57.7 to 73.2]

16. Secondary Outcome: Antibody Concentrations for Anti-PT, Anti-FHA and Anti-PRN, Post Booster Vaccination
Description: The antibody concentrations for anti-PT, anti-FHA and anti-PRN were presented as GMCs and expressed as IU/mL.
Time Frame: At Month 16 (i.e. one month after booster vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 188
IU/mL
  anti-FHA antibody | 268.4 [242.4 to 297.2]
  anti-PRN antibody: number analyzed (Participants) | 187
  anti-PRN antibody | 563.4 [495.6 to 640.5]
  anti-PT antibody | 107.9 [96.5 to 120.7]

17. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs) Following Each Dose of Primary Vaccination
Description: The solicited local AEs assessed were pain, redness and swelling at injection site. Any = Occurrence of the AE regardless of the intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after each primary vaccination dose (i.e. at Day 0, at Month 1.5 and at Month 3)
Population: Total vaccinated cohort (TVC) for analysis of safety of the primary epoch: all subjects with at least one primary vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 232
Participants
  Any Pain, Dose 1 | 58
  Any Redness, Dose 1 | 83
  Any Swelling, Dose 1 | 45
  Any Pain, Dose 2: number analyzed (Participants) | 229
  Any Pain, Dose 2 | 47
  Any Redness, Dose 2: number analyzed (Participants) | 229
  Any Redness, Dose 2 | 89
  Any Swelling, Dose 2: number analyzed (Participants) | 229
  Any Swelling, Dose 2 | 58
  Any Pain, Dose 3: number analyzed (Participants) | 226
  Any Pain, Dose 3 | 50
  Any Redness, Dose 3: number analyzed (Participants) | 226
  Any Redness, Dose 3 | 96
  Any Swelling, Dose 3: number analyzed (Participants) | 226
  Any Swelling, Dose 3 | 63

18. Secondary Outcome: Number of Subjects With Any Solicited Local AEs Following Booster Vaccination
Description: as for outcome 17
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination dose (i.e. at Month 15)
Population: Total vaccinated cohort (TVC) for analysis of safety of the booster epoch: all subjects with at least one booster vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 225
Participants
  Any Pain | 71
  Any Redness | 101
  Any Swelling | 73

19. Secondary Outcome: Number of Subjects With Any Solicited General AEs Following Each Dose of Primary Vaccination
Description: The solicited general AEs assessed were drowsiness, irritability/fussiness, loss of appetite and fever. Any = Occurrence of the AE regardless of the intensity grade. Any fever = Fever (axillary) ≥ 37.5°C.
Time Frame: as for outcome 17
Population: TVC for analysis of safety of the primary epoch: all subjects with at least one primary vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 232
Participants
  Any Drowsiness, Dose 1 | 82
  Any Irritability / Fussiness, Dose 1 | 100
  Any Loss Of Appetite, Dose 1 | 33
  Any Temperature/(Axillary) (°C), Dose 1 | 14
  Any Drowsiness, Dose 2: number analyzed (Participants) | 230
  Any Drowsiness, Dose 2 | 69
  Any Irritability / Fussiness, Dose 2: number analyzed (Participants) | 230
  Any Irritability / Fussiness, Dose 2 | 104
  Any Loss Of Appetite, Dose 2: number analyzed (Participants) | 230
  Any Loss Of Appetite, Dose 2 | 34
  Any Temperature/(Axillary) (°C), Dose 2: number analyzed (Participants) | 230
  Any Temperature/(Axillary) (°C), Dose 2 | 32
  Any Drowsiness, Dose 3: number analyzed (Participants) | 225
  Any Drowsiness, Dose 3 | 65
  Any Irritability / Fussiness, Dose 3: number analyzed (Participants) | 225
  Any Irritability / Fussiness, Dose 3 | 106
  Any Loss Of Appetite, Dose 3: number analyzed (Participants) | 225
  Any Loss Of Appetite, Dose 3 | 43
  Any Temperature/(Axillary) (°C), Dose 3: number analyzed (Participants) | 225
  Any Temperature/(Axillary) (°C), Dose 3 | 28

20. Secondary Outcome: Number of Subjects With Any Solicited General AEs Following Booster Vaccination
Description: as for outcome 19
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination dose (i.e. at Month 15)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 225
Participants
  Any Drowsiness | 54
  Any Irritability / Fussiness | 88
  Any Loss Of Appetite | 40
  Any Temperature/(Axillary) (°C) | 26

21. Secondary Outcome: Number of Subjects With Unsolicited AEs Following Each Dose of Primary Vaccination
Description: An unsolicited AE was defined as any AE reported in addition to those solicited during the clinical study and any solicited AE with onset outside the specified period of follow-up for solicited AEs. Any = Occurrence of the AE regardless of the intensity grade.
Time Frame: During the 31-day (Days 0-30) follow-up period after each primary vaccination dose (i.e. at Day 0, at Month 1.5 and at Month 3)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 235
Participants | 48

22. Secondary Outcome: Number of Subjects With Unsolicited AEs Following Booster Vaccination
Description: as for outcome 21
Time Frame: During the 31-day (Days 0-30) follow-up period after booster vaccination dose (i.e. at Month 15)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 225
Participants | 13

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: The SAEs assessed included any untoward medical occurrences that resulted in death, were life threatening, required hospitalisation or prolongation of existing hospitalisation or resulted in disability/incapacity. Any = Occurrence of the AE regardless of the intensity grade.
Time Frame: During the entire study period (i.e. from Day 0 until Month 16)
Population: TVC for analysis of safety of the primary epoch: all subjects with at least one primary vaccine dose administration documented, and TVC for analysis of safety of the booster epoch: all subjects with the booster vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | DTPa-IPV/Hib Group
Number analyzed (Participants) | 235
Participants | 3

ADVERSE EVENTS:
Time Frame: Solicited local & general AEs: during the 4-day (Days 0-3) follow-up period after each primary & booster vaccination. Unsolicited AEs: during the 31-day (Days 0-30) follow-up period after each primary & booster vaccination. SAEs: from Day 0 until Month 16.
Description: Solicited local and general AEs, unsolicited AEs, and SAEs were reported for the Primary Epoch and for the Booster Epoch.
Arm/Group | DTPa-IPV/Hib Group
All-Cause Mortality (participants affected / at risk) | 0/235
Serious Adverse Events (participants affected / at risk) | 3/235
Other Adverse Events (participants affected / at risk) | 201/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTPa-IPV/Hib Group (N=235)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTPa-IPV/Hib Group (N=235)
Agitation (Psychiatric disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Cardiovascular disorder (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 93 (150)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (2)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 1 (2)
Injection site erythema (General disorders) | 140 (369)
Injection site pain (General disorders) | 103 (226)
Injection site swelling (General disorders) | 102 (239)
Nightmare (Psychiatric disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2)
Poor quality sleep (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 67 (104)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 5 (6)
Rhinitis (Infections and infestations) | 15 (18)
Somnolence (Nervous system disorders) | 131 (270)
Tracheitis (Infections and infestations) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (7)
Urinary tract infection (Infections and infestations) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Varicella (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Irritability postvaccinal (General disorders) | 157 (398)
Enteritis infectious (Infections and infestations) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02858440/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT02858440/SAP_001.pdf